CLINICAL TRIAL: NCT02357394
Title: Cervical Pessary to Prevent Preterm Birth in Singleton Pregnancies With a Sonographically Measured Short Cervix: an Open-label Randomized Controlled Trial
Brief Title: Cervical Pessary to Prevent Preterm Birth in Singleton Pregnancies With a Sonographically Measured Short Cervix
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit patients
Sponsor: Gene Lee, MD (Other)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor-Investigator, Gene Lee, MD, Assistant Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUOBGYN001
Record Dates: First submitted 2015-01-13; First posted 2015-02-06 (Estimated); Results first posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Premature Birth
Keywords: arabin pessary; short cervix
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Device: Arabin Pessary (Experimental): Participants randomized to this group will receive the pessary.
  Interventions: Device: Arabin Pessary
- Standard of Care (No Intervention): Patients randomized to the control group will receive standard of care for their condition. This includes surveillance of cervical length, vaginal progesterone, and emergency cerclage.

INTERVENTIONS:
Device: Arabin Pessary — Arabin pessary is a ring manufactured from medical grade silicone. It comes in 13 different sizes. Participants will be fitted to the appropriate size by the study team.
  Arms: Device: Arabin Pessary

SUMMARY:
The purpose of this study is to learn if the Arabin pessary can reduce preterm birth less than 37 weeks 0 days in singleton pregnancies that have a short cervix.

DETAILED DESCRIPTION:
This is an open label randomized controlled study. The pessary will be offered to those patients who have a transvaginal cervical length less than 25 mm before 23 weeks 0 days. The control group will receive the current standard of care which includes surveillance of cervical length, vaginal progesterone, and emergency cerclage. The primary outcome of the study is preterm delivery less than 37 weeks 0 days.

ELIGIBILITY:
Inclusion Criteria:

* singleton
* cervical length < 25 mm measured by transvaginal ultrasound prior to 23 weeks 0 days
* agrees to refrain from sexual intercourse

Exclusion Criteria:

* major fetal anomalies
* painful regular uterine contractions
* active vaginal bleeding
* ruptured membranes
* evidence of chorioamnionitis or other maternal/fetal infectious morbidity
* placenta previa
* cervical cerclage in situ
* visual cervical dilation of 2 cm or greater with visible amnion/chorion
* significant maternal-fetal complications (chronic hypertension, insulin dependent diabetes mellitus, systemic lupus erythematosus with nephritis, chronic hypertension, red cell alloimmunization, drug abuse)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2015-05; Primary Completion 2017-06-06 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gene T Lee, MD, Principal Investigator — University of Kansas Medical Center; Eugene Y Chang, MD, Principal Investigator — Medical University of South Carolina; Carl P Weiner, MD, MBA, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Participating in GoNet IPD of pessary for prevention of preterm birth.

REFERENCES:
- [Background] Carreras E, Arevalo S, Bello-Munoz JC, Goya M, Rodo C, Sanchez-Duran MA, Peiro JL, Cabero L. Arabin cervical pessary to prevent preterm birth in severe twin-to-twin transfusion syndrome treated by laser surgery. Prenat Diagn. 2012 Dec;32(12):1181-5. doi: 10.1002/pd.3982. Epub 2012 Oct 11. PMID 23055333
- [Background] Goya M, Pratcorona L, Merced C, Rodo C, Valle L, Romero A, Juan M, Rodriguez A, Munoz B, Santacruz B, Bello-Munoz JC, Llurba E, Higueras T, Cabero L, Carreras E; Pesario Cervical para Evitar Prematuridad (PECEP) Trial Group. Cervical pessary in pregnant women with a short cervix (PECEP): an open-label randomised controlled trial. Lancet. 2012 May 12;379(9828):1800-6. doi: 10.1016/S0140-6736(12)60030-0. Epub 2012 Apr 3. PMID 22475493
- [Background] Ting YH, Lao TT, Wa Law L, Hui SY, Chor CM, Lau TK, Yeung Leung T. Arabin cerclage pessary in the management of cervical insufficiency. J Matern Fetal Neonatal Med. 2012 Dec;25(12):2693-5. doi: 10.3109/14767058.2012.712559. Epub 2012 Aug 22. PMID 22871155
- [Background] Sieroszewski P, Jasinski A, Perenc M, Banach R, Oszukowski P. The Arabin pessary for the treatment of threatened mid-trimester miscarriage or premature labour and miscarriage: a case series. J Matern Fetal Neonatal Med. 2009 Jun;22(6):469-72. doi: 10.1080/14767050802531748. PMID 19530009
- [Background] Arabin B, Halbesma JR, Vork F, Hubener M, van Eyck J. Is treatment with vaginal pessaries an option in patients with a sonographically detected short cervix? J Perinat Med. 2003;31(2):122-33. doi: 10.1515/JPM.2003.017. PMID 12747228
- [Background] Quaas L, Hillemanns HG, du Bois A, Schillinger H. [The Arabin cerclage pessary--an alternative to surgical cerclage]. Geburtshilfe Frauenheilkd. 1990 Jun;50(6):429-33. doi: 10.1055/s-2008-1026276. German. PMID 2198191
- [Background] Liem S, Schuit E, Hegeman M, Bais J, de Boer K, Bloemenkamp K, Brons J, Duvekot H, Bijvank BN, Franssen M, Gaugler I, de Graaf I, Oudijk M, Papatsonis D, Pernet P, Porath M, Scheepers L, Sikkema M, Sporken J, Visser H, van Wijngaarden W, Woiski M, van Pampus M, Mol BW, Bekedam D. Cervical pessaries for prevention of preterm birth in women with a multiple pregnancy (ProTWIN): a multicentre, open-label randomised controlled trial. Lancet. 2013 Oct 19;382(9901):1341-9. doi: 10.1016/S0140-6736(13)61408-7. Epub 2013 Aug 5. PMID 23924878
- [Background] Liem SM, van Baaren GJ, Delemarre FM, Evers IM, Kleiverda G, van Loon AJ, Langenveld J, Schuitemaker N, Sikkema JM, Opmeer BC, van Pampus MG, Mol BW, Bekedam DJ. Economic analysis of use of pessary to prevent preterm birth in women with multiple pregnancy (ProTWIN trial). Ultrasound Obstet Gynecol. 2014 Sep;44(3):338-45. doi: 10.1002/uog.13432. Epub 2014 Aug 7. PMID 24898103

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Device: Arabin Pessary | Standard of Care
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Device: Arabin Pessary | Standard of Care | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Full Range); unit: years] | 37.2 [25 to 44] | 36 [31 to 39] | 36.7 [25 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7
marital status [Count of Participants; unit: Participants]
  married or living with partner | 3 | 3 | 6
  never married | 1 | 0 | 1
employment status [Count of Participants; unit: Participants]
  full time | 2 | 3 | 5
  unemployed | 1 | 0 | 1
  part-time | 1 | 0 | 1
years education [Mean (Full Range); unit: years] — Population: missing data
  years
    number analyzed (Participants) | 4 | 1 | 5
    (all) | 14.5 [12 to 18] | 14 [14 to 14] | 14.4 [12 to 18]
insurance group [Count of Participants; unit: Participants]
  private insurance | 4 | 3 | 7
  uninsured | 0 | 0 | 0
  government insurance | 0 | 0 | 0
tobacco use [Count of Participants; unit: Participants] | 1 | 0 | 1
alcohol use [Count of Participants; unit: Participants] | 0 | 0 | 0
prepreg BMI [Mean (Full Range); unit: kg/m^2] | 22.4 [19.6 to 25.4] | 36.4 [31.8 to 39.9] | 28.4 [19.6 to 39.9]
infections before enrollment [Count of Participants; unit: Participants] | 0 | 0 | 0
infections at enrollment [Count of Participants; unit: Participants] | 1 | 0 | 1
nullipara [Count of Participants; unit: Participants] | 0 | 1 | 1
# of pregnancies < 16 wk delivered spontaneously [Mean (Full Range); unit: pregnancies] | 0.25 [0 to 1] | 1 [0 to 2] | 0.6 [0 to 2]
# of pregnancies 16w0d-23w6d delivered spontaneously [Mean (Full Range); unit: pregnancies] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
# of pregnancies 24w0d-36w6d delivered sponaneously [Mean (Full Range); unit: pregnancies] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
prior operative vaginal delivery [Count of Participants; unit: Participants]
  yes | 1 | 0 | 1
  no | 3 | 3 | 6
prior Cesarean [Count of Participants; unit: Participants]
  yes | 1 | 0 | 1
  no | 3 | 3 | 6
prior cervical surgery [Count of Participants; unit: Participants]
  yes | 0 | 0 | 0
  no | 4 | 3 | 7
gestational weeks at randomization [Mean (Full Range); unit: weeks] | 21.4 [20.1 to 22.6] | 19.6 [17.4 to 21.2] | 20.7 [17.4 to 22.6]
TVCL at randomization [Mean (Full Range); unit: millimeters] | 15.8 [10.2 to 20.8] | 20.2 [17 to 22] | 17.7 [10.2 to 22]
Funneling present [Count of Participants; unit: Participants] | 4 | 2 | 6
sludge present [Count of Participants; unit: Participants] | 2 | 0 | 2
progesterone started? [Count of Participants; unit: Participants] | 0 | 2 | 2
cerclage placed? [Count of Participants; unit: Participants] | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Preterm Birth Before 37 Weeks
Description: Preterm birth refers to pregnancies that deliver before 37 weeks. Count of participants that deliver before they reach 37 weeks.
Time Frame: Up to 37 weeks 0 days
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Arabin Pessary | Standard of Care
Number analyzed (Participants) | 4 | 3
Participants | 3 | 1

2. Secondary Outcome: Preterm Birth Before 34 Weeks
Description: Number of deliveries before 34 weeks 0 days of gestation
Time Frame: up to 34 weeks 0 days
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Arabin Pessary | Standard of Care
Number analyzed (Participants) | 4 | 3
Participants | 1 | 0

3. Secondary Outcome: Neonatal Composite Morbidity
Description: Count of Fetal or Neonatal death up to 28 days after birth, respiratory distress syndrome, chronic lung disease, periventricular lucency, periventricular leukomalacia, intraventricular hemorrhage grade 3 or 4, necrotizing enterocolitis, early-onset-culture-proven sepsis
Time Frame: antepartum and up to 28 days after postnatal gestational age of 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Arabin Pessary | Standard of Care
Number analyzed (Participants) | 4 | 3
Participants | 1 | 0

4. Secondary Outcome: Neonatal Length of Stay
Description: Total number of days in hospital after birth
Time Frame: participants will be followed for the duration of hospital stay, up to 17 weeks after delivery
Measure: Mean (Full Range); unit: days
Arm/Group | Device: Arabin Pessary | Standard of Care
Number analyzed (Participants) | 3 | 3
days | 3.3 [3 to 4] | 7 [2 to 16]

5. Secondary Outcome: Admission to Neonatal Intensive Care Unit
Description: Number of babies admitted to neonatal intensive care unit after birth during the same hospital stay.
Time Frame: participants will be followed for the duration of hospital stay, up to 17 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Arabin Pessary | Standard of Care
Number analyzed (Participants) | 3 | 3
Participants | 0 | 1

6. Secondary Outcome: Total Days in the Neonatal Intensive Care Unit
Description: Number of days a baby spends in the neonatal intensive care unit
Time Frame: participants will be followed for the duration of hospital stay, up to 17 weeks after delivery
Measure: Mean (Full Range); unit: days
Arm/Group | Device: Arabin Pessary | Standard of Care
Number analyzed (Participants) | 3 | 3
days | 0 [0 to 0] | 16 [16 to 16]

7. Secondary Outcome: Duration of Ventilator Support
Description: Number of days a baby requires use of mechanical ventilation
Time Frame: participants will be followed for the duration of hospital stay, up to 17 weeks after delivery
Measure: Mean (Full Range); unit: days
Arm/Group | Device: Arabin Pessary | Standard of Care
Number analyzed (Participants) | 3 | 3
days | 0 [0 to 0] | 0 [0 to 0]

8. Secondary Outcome: Retinopathy of Prematurity Requiring Treatment
Description: Number of newborn with Retinopathy of Prematurity that requires intervention.
Time Frame: participants will be followed for the duration of hospital stay, up to 17 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Arabin Pessary | Standard of Care
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

9. Secondary Outcome: Birthweight < 1500 Grams
Description: Number of newborns whose birthweight is less than 1500 grams
Time Frame: at time of birth, expected to be within 4 weeks of due date
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Arabin Pessary | Standard of Care
Number analyzed (Participants) | 4 | 3
Participants | 1 | 0

10. Secondary Outcome: Birthweight < 2500 Grams
Description: Number of newborns whose birthweight is less than 2500 grams
Time Frame: at time of birth, expected to be within 4 weeks of due date
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Arabin Pessary | Standard of Care
Number analyzed (Participants) | 4 | 3
Participants | 3 | 1

11. Secondary Outcome: Gestational Age at Delivery
Description: Number of weeks of gestation completed by time of delivery
Time Frame: at time of birth, expected to be within 4 weeks of due date
Measure: Mean (Full Range); unit: weeks
Arm/Group | Device: Arabin Pessary | Standard of Care
Number analyzed (Participants) | 4 | 3
weeks | 33.1 [21.1 to 39] | 37.3 [34 to 39.4]

12. Secondary Outcome: Use of Tocolysis
Description: Number of participants required use of tocolytic medication
Time Frame: participants will be followed for the duration of pregnancy, up to nine months
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Arabin Pessary | Standard of Care
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

13. Secondary Outcome: Use of Antenatal Steroids
Description: Number of participants that received betamethasone or dexamethasone to reduce morbidity of expected preterm delivery
Time Frame: participants will be followed for the duration of pregnancy, up to nine months
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Arabin Pessary | Standard of Care
Number analyzed (Participants) | 4 | 3
Participants | 0 | 3

14. Secondary Outcome: Chorioamnionitis
Description: Number of participants that showed intrauterine infection diagnosed by maternal tachycardia, fever, uterine tenderness, purulent or abnormal cervical discharge, fetal tachycardia.
Time Frame: participants will be followed for the duration of pregnancy, up to nine months
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Arabin Pessary | Standard of Care
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

15. Secondary Outcome: Vaginal Bleeding
Description: Number of participants who experienced bleeding from lower genital tract during antepartum period
Time Frame: participants will be followed for the duration of pregnancy, up to nine months
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Arabin Pessary | Standard of Care
Number analyzed (Participants) | 4 | 3
Participants | 1 | 0

16. Secondary Outcome: Preterm Premature Rupture of Membranes
Description: Number of participants who experienced rupture of membranes as diagnosed by speculum exam showing pooling, ferning, positive nitrazine test, positive amnisure test.
Time Frame: participants will be followed for the duration of pregnancy, up to nine months
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Arabin Pessary | Standard of Care
Number analyzed (Participants) | 4 | 3
Participants | 1 | 1

17. Secondary Outcome: Cesarean Delivery
Description: Number of participants that underwent cesarean delivery
Time Frame: at time of delivery, expected to be within 4 weeks of due date
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Arabin Pessary | Standard of Care
Number analyzed (Participants) | 4 | 3
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 year, 5 months
Arm/Group | Device: Arabin Pessary | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

LIMITATIONS AND CAVEATS:
Study closed due to poor enrollment, unable to complete.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT02357394/Prot_SAP_000.pdf